CLINICAL TRIAL: NCT01244815
Title: Efficacy and Safety of 3-Week Fixed-Dose Asenapine Treatment in Pediatric Acute Manic or Mixed Episodes Associated With Bipolar I Disorder (Protocol No. P06107)
Brief Title: Efficacy and Safety of Asenapine Treatment for Pediatric Bipolar Disorder (P06107 Has an Extension [P05898; NCT01349907])(P06107)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06107
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2022-02

CONDITIONS: Bipolar Disorder, Pediatric
Keywords: Bi-polar I disorder; antipsychotic; serotonin; dopamine; noradrenalin; histamine; pediatric
MeSH Terms: conditions — Bipolar Disorder | interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Asenapine 2.5 mg twice daily (BID) (Experimental): Participants receive asenapine 2.5 mg BID for 21 days.
  Interventions: Drug: asenapine; Drug: Rescue medication
- Asenapine 5.0 mg BID (Experimental): Participants receive asenapine 2.5 mg BID through Day 3. On Day 4 participants receive asenapine 2.5 mg in the morning and 5.0 mg in the evening. Participants receive asenapine 5.0 mg BID for the remainder of the 21-day treatment period.
  Interventions: Drug: asenapine; Drug: Rescue medication
- Asenapine 10.0 mg BID (Experimental): Participants receive asenapine 2.5 mg BID through Day 3. On Day 4 participants receive asenapine 2.5 mg in the morning and 5.0 mg in the evening. On Day 5 and 6 participants receive asenapine 5.0 mg BID. On Day 7 participants receive asenapine 5.0 mg in the morning and 10.0 mg in the evening. Participants receive asenapine 10.0 mg BID for the remainder of the 21-day treatment period.
  Interventions: Drug: asenapine; Drug: Rescue medication
- Placebo (Placebo Comparator): Participants receive placebo BID for 21 days.
  Interventions: Drug: Placebo to match asenapine; Drug: Rescue medication

INTERVENTIONS:
Drug: asenapine — Asenapine tablets, administered sublingually twice daily at one of three dose levels (2.5 mg, 5.0 mg, or 10.0 mg)
  Other Names: SCH 900274, Saphris
  Arms: Asenapine 10.0 mg BID; Asenapine 2.5 mg twice daily (BID); Asenapine 5.0 mg BID
Drug: Placebo to match asenapine — Placebo tablets to match asenapine tablets, administered sublingually twice daily
  Arms: Placebo
Drug: Rescue medication — For participants whose symptoms worsen or are not adequately controlled on assigned treatment, rescue medication may be administered during the trial in the following circumstances. For the control of agitation, anxiety, insomnia, restlessness, or akathisia and extrapyramidal symptoms (EPS) some benzodiazepines and EPS medications (i.e., anticholinergics) are allowed. Benadryl (diphenhydramine) and beta blockers are also permitted, provided that they are not taken within 8 hours of efficacy assessments.

SUMMARY:
Efficacy and safety of asenapine for the treatment of bipolar I disorder (manic or mixed episodes) will be evaluated in participants between 10 and 17 years old, who are either hospitalized or non-hospitalized. In this 3-weeks, double-blind, parallel design trial, eligible participants will be randomized to receive one out of three fixed dose levels of asenapine, or placebo. The study primary hypothesis is that at least one asenapine dose is superior to placebo as measured by the change from baseline to Day 21 in Young Mania Rating Scale (Y-MRS) total score. Trial medication and placebo are provided as identical-looking sublingual tablets; concurrent use of psychotropics is prohibited, except use of short-acting benzodiazepines and psychostimulants approved for the treatment of attention deficit hyperactivity disorder (ADHD). Main treatment effect is measured using Y-MRS and safety is evaluated using the recordings of adverse events, routine blood panels, physical examinations (including vital signs), and electrocardiograms. Participants who complete the double blind trial may be offered to continue (open-label) treatment with asenapine for an extended period of time. Follow-up information on safety parameters will be collected in all participants within 30 days following treatment discontinuation.

DETAILED DESCRIPTION:
Participants' Y-MRS total score at baseline will be subtracted from that at the Day 21 visit to determine the amount of change over time with treatment. The responses for the 3 different asenapine doses compared to placebo will be evaluated. The Y-MRS is an 11 item scale: seven items ranked on scale from 0 to 4 and four items ranked 0 to 8 with a range of possible total scores from 0 to 60.

Participants' overall score on the CGI-BP at Day 21 will be evaluated to determine the amount of change over time with treatment. The responses for the 3 different asenapine doses compared to placebo will be evaluated. CGI-BP overall score is obtained from a single-item clinician-rated scale used to assess the participant's overall bipolar illness. Scores range from not ill (1) to very severely ill (7).

The proportion of participants whose total Y-MRS score is decreased ≥50% from baseline at Day 4, 7, 14 and 21. Results for the 3 different asenapine doses compared to placebo will be evaluated.

Participants' mania sub-score from the CGI-BP will be evaluated for each study visit (Days 4, 7, 14 and 21) to determine the amount of change over time with treatment. The responses for the 3 different asenapine doses compared to placebo will be evaluated.

Participants' depression sub-score from the CGI-BP will evaluated at each study visit (Days 4, 7, 14 and 21) to determine the amount of change over time with treatment. The responses for the 3 different asenapine doses compared to placebo will be evaluated.

Participants' CDRS-R at baseline will be subtracted from those at each study visit at which this rating was measured (Days 7, 14 and 21) to determine the amount of change over time with treatment. The responses for the 3 different asenapine doses compared to placebo will be evaluated. The CDRS-R is a 17-item scale that assesses the presence and severity of depressive symptoms: fourteen items are rated from 1 to 7 and three items are rated from 1 to 5; total scores range from 17 to 113.

Participants' CGAS at baseline will be subtracted from that at the Day 21 visit to determine the amount of change over time with treatment. The responses for the 3 different asenapine doses compared to placebo will be evaluated. The CGAS is a 100-point scale, with a possible range of 1 to 100. Normal social functioning is defined as a CGAS total score of ≥70.

Participants' PQ-LES-Q total score at baseline will be subtracted from that at the Day 21 visit to determine the amount of change over time with treatment. The responses for the 3 different asenapine doses compared to placebo will be evaluated. The PQ-LES-Q is a 15-item scale, with total score calculated as the sum of the first 14 items, with a range of 14 to 70. Each item is scored by the child from 1 to 5, with higher scores indicative of greater enjoyment and satisfaction.

Participants' PQ-LES-Q overall score (i.e. item 15) at baseline will be subtracted from that at the Day 21 visit to determine the amount of change over time with treatment. The responses for the 3 different asenapine doses compared to placebo will be evaluated. The PQ-LES-Q overall score is determined by the answer to item 15 on the questionnaire (range: 1 to 5).

ELIGIBILITY:
Inclusion criteria:

* Participants who (or whose parent/legal representative) are able to give written informed consent.
* Participants must be 10 years of age or older and 17 years of age or younger at the time of treatment assignment (randomization).
* Participants must have a diagnosis of bipolar I disorder, confirmed by structured interview at screening.
* Participants must not be pregnant or lactating, and those who are sexually active or become sexually active during the trial, and of child-bearing potential, must be using a medically accepted form of birth control.
* Participants will be required to have stopped taking certain psycho-active medications prior to baseline.
* Participants must have a caregiver, or other responsible person living with them who agrees to provide support to the participant to ensure study and procedure compliance.

Exclusion criteria:

* Diagnosis of bipolar II disorder, or other form of bipolar or psychotic disorder.
* Known or suspected mental retardation.
* Substance abuse, or dependence, within the past 6 months.
* There is risk of self-harm or harm to others.
* There is a history of tardive dyskinesia or dystonia.
* Pregnancy or lactation during the study.
* History of seizure disorder.
* Participation in any other clinical trial at the same time.
* A family member who is part of the study staff or is directly involved with the study.
* Other medical conditions determined by the study staff to possibly interfere with the study safety and efficacy evaluations.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 404 (Actual)
Dates: Start 2011-06-16 (Actual); Primary Completion 2013-08-28 (Actual); Study Completion 2013-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Findling RL, Landbloom RL, Szegedi A, Koppenhaver J, Braat S, Zhu Q, Mackle M, Chang K, Mathews M. Asenapine for the Acute Treatment of Pediatric Manic or Mixed Episode of Bipolar I Disorder. J Am Acad Child Adolesc Psychiatry. 2015 Dec;54(12):1032-41. doi: 10.1016/j.jaac.2015.09.007. Epub 2015 Oct 24. PMID 26598478

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants receive placebo twice daily (BID) for 21 days.
- Asenapine 2.5 mg BID: Participants receive asenapine 2.5 mg BID for 21 days.
Period: Overall Study
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Started | 101 (Randomized) | 105 (Randomized) | 99 (Randomized) | 99 (Randomized)
Treated | 101 | 104 | 99 | 99
Completed | 87 | 88 | 88 | 87
Not Completed | 14 | 17 | 11 | 12
Not completed — Not Treated | 0 | 1 | 0 | 0
Not completed — Adverse Event | 4 | 7 | 5 | 5
Not completed — Treatment Failure | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 3 | 2 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 3
Not completed — Protocol Violation | 7 | 4 | 3 | 1
Not completed — Did Not Meet Protocol Eligibility | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The population consisted of all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID | Total
Number analyzed (Participants) | 101 | 104 | 99 | 99 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (2.0) | 13.7 (2.1) | 13.8 (2.0) | 13.9 (2.1) | 13.8 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 52 | 56 | 41 | 212
  Male | 38 | 52 | 43 | 58 | 191
Young Mania Rating Scale (Y-MRS) total score [Mean (Standard Deviation); unit: score on a scale] — Y-MRS is an 11-item instrument for assessing the severity of manic episodes. Seven of the 11 items are rated on a scale of 0-4 and 4 are rated on a scale of 0-8, with higher scores indicating greater severity of symptoms. The Y-MRS total score for each participant is the sum of the ratings for the 11 individual items, and can range from 0-60. Summary statistics presented are for efficacy population (Full Analysis Set [FAS]): N=98, 101, 98, 98 and 395 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID, asenapine 10.0 mg BID and Total groups, respectively.
  score on a scale | 29.9 (5.5) | 29.5 (5.7) | 30.3 (5.9) | 30.2 (5.6) | 30.0 (5.7)
Clinical Global Impression Scale for use in Bipolar Disorder (CGI-BP) overall score [Mean (Standard Deviation); unit: score on a scale] — CGI-BP overall score is obtained using a 7-point scale assessing the severity of the participant's overall bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. Summary statistics presented are for efficacy population (FAS): N=98, 101, 98, 98 and 395 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID, asenapine 10.0 mg BID and Total groups, respectively.
  score on a scale | 4.3 (0.5) | 4.5 (0.6) | 4.4 (0.6) | 4.4 (0.6) | 4.4 (0.6)
CGI-BP mania score [Mean (Standard Deviation); unit: score on a scale] — CGI-BP mania score is obtained using a 7-point scale assessing the severity of the mania component of the participant's bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. Summary statistics presented are for efficacy population (FAS): N=98, 101, 98, 98 and 395 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID, asenapine 10.0 mg BID and Total groups, respectively.
  score on a scale | 4.3 (0.5) | 4.5 (0.6) | 4.4 (0.6) | 4.4 (0.6) | 4.4 (0.6)
CGI-BP depression score [Mean (Standard Deviation); unit: score on a scale] — CGI-BP depression score is obtained using a 7-point scale assessing the severity of the depression component of the participant's bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. Summary statistics presented are for efficacy population (FAS) except as noted: N=97 (baseline value not available for 1 FAS participant in this group), 101, 98, 98 and 394 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID, asenapine 10.0 mg BID and Total groups, respectively.
  score on a scale | 2.9 (1.3) | 2.8 (1.3) | 2.9 (1.4) | 2.8 (1.2) | 2.8 (1.3)
Children's Depression Rating Scale, Revised (CDRS-R) total score [Mean (Standard Deviation); unit: score on a scale] — CDRS-R is a 17-item instrument for assessing depression in children. Items are rated on a scale of 1-7 (14 items) or 1-5 (3 items); higher scores indicate more severe symptoms. CDRS-R total score is sum of ratings for the 17 items (range: 17-113). Summary statistics presented are for efficacy population (FAS) except as noted: N=97 (baseline value not available for 1 FAS participant in this group), 99 (baseline value not available for 2 FAS participants in this group), 98, 98 and 392 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID, asenapine 10.0 mg BID and Total groups, respectively.
  score on a scale | 34.5 (10.2) | 33.7 (9.0) | 35.2 (11.9) | 34.1 (9.0) | 34.4 (10.1)
Children's Global Assessment Scale (CGAS) total score - current functioning [Mean (Standard Deviation); unit: score on a scale] — CGAS is a 100-point scale measuring psychological, social, and school functioning in children aged 6-17. Minimum scores ranged from 1-10, representing the need for constant supervision (worse result) to maximum scores of 91-100, representing superior functioning (better result). Summary statistics presented are for efficacy population (Full Analysis Set [FAS]): N=98, 101, 98, 98 and 395 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID, asenapine 10.0 mg BID and Total groups, respectively.
  score on a scale | 49.0 (7.9) | 49.6 (7.4) | 48.4 (7.4) | 49.1 (6.7) | 49.0 (7.4)
Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) total score [Mean (Standard Deviation); unit: score on a scale] — PQ-LES-Q is a questionnaire to assess quality of life enjoyment and satisfaction in children and adolescents. The participant is asked to rate 15 items reflecting quality of life on a scale of 1=very poor to 5=very good. The PQ-LES-Q total score (sum of Items 1-14) ranged from 14 to 70 with a higher score indicating better quality of life. Summary statistics presented are for efficacy population (Full Analysis Set [FAS]): N=98, 101, 98, 98 and 395 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID, asenapine 10.0 mg BID and Total groups, respectively.
  score on a scale | 48.7 (9.7) | 49.1 (9.6) | 49.5 (9.1) | 49.1 (10.5) | 49.1 (9.7)
PQ-LES-Q overall score (i.e., item 15) [Mean (Standard Deviation); unit: score on a scale] — PQ-LES-Q is a questionnaire to assess quality of life enjoyment and satisfaction in children and adolescents. The participant is asked to rate 15 items reflecting quality of life on a scale of 1=very poor to 5=very good. The PQ-LES-Q overall score (Item 15, a global assessment of quality of life) ranged from 1 to 5 with a higher score indicating better quality of life. Summary statistics presented are for efficacy population (Full Analysis Set [FAS]): N=98, 101, 98, 98 and 395 for Placebo, asenapine 2.5 mg BID, asenapine 5.0 mg BID, asenapine 10.0 mg BID and Total groups, respectively.
  score on a scale | 3.7 (1.0) | 3.8 (1.0) | 3.8 (0.9) | 3.8 (1.0) | 3.8 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Y-MRS Total Score at Day 21
Description: The Y-MRS is an 11-item clinician-rated instrument for assessing the severity of manic episodes. A severity rating is assigned to each of the 11 items (Elevated mood, Increased motor activity-energy, Sexual interest, Sleep, Irritability, Speech, Language-thought disorder, Thought content, Disruptive-aggressive behavior, Appearance, Insight), based on the participant's subjective report of his or her condition over the previous 48 hours and the clinician's observations during the interview, with the emphasis on the latter. Seven of the 11 items are rated on a scale of 0-4 and 4 of the items are rated on a scale of 0-8, with higher scores indicating greater severity of symptoms. The Y-MRS total score for each participant is the sum of the ratings for the 11 individual items, and can range from 0-60, with higher scores indicating greater severity of symptoms. The reported measure is the change from baseline at Day 21; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 21
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy Full Analysis Set [FAS]); also, to be included an on-treatment Day 21 value of Y-MRS total score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 79 | 88 | 87 | 81
score on a scale | -9.6 (7.8) | -12.3 (9.0) | -15.1 (9.5) | -15.9 (9.1)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Model uses efficacy FAS population (number of participants: placebo - 98, asenapine 2.5 mg - 101, asenapine 5.0 mg - 98, asenapine 10.0 mg - 98); Test type: Superiority or Other; p = 0.008, Mixed Model for Repeated Measures (MMRM) — p-value is adjusted by Hochberg's method for testing three asenapine groups versus the placebo group; Model included terms of (pooled) site, treatment, visit, baseline, and the interaction of visit by treatment and baseline by visit; Difference in Least Squares (LS) Means = -3.2, 95% CI 2-sided [-5.6 to -0.8] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM — p-value is adjusted by Hochberg's method for testing three asenapine groups versus the placebo group; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -5.3, 95% CI 2-sided [-7.7 to -2.9] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM — p-value is adjusted by Hochberg's method for testing three asenapine groups versus the placebo group; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -6.2, 95% CI 2-sided [-8.6 to -3.8] — Estimate is asenapine versus placebo
Statistical Analysis 4: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID vs Asenapine 10.0 mg BID; Investigation of dose-response relationship of change from baseline to Day 21 in Y-MRS total score was a Secondary study endpoint. Multiple contrast testing using MMRM model (FAS population) was used to evaluate 7 pre-defined dose-response patterns; Test type: Superiority or Other; p < 0.0001, MMRM — p-value (adjusted to control Type I error in multiple testing) for dose-response pattern 1 (Placebo<2.5 mg=5.0 mg=10.0 mg); [statistical method as in outcome 1, analysis 1]; t-statistic = -4.92 — t-statistic associated with the contrast of the MMRM model for dose-response pattern 1. Lower value indicates pattern provides better fit to data
Statistical Analysis 5: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.0001, MMRM — p-value (adjusted to control Type I error in multiple testing) for dose-response pattern 2 (Placebo=2.5 mg<5.0 mg=10.0 mg); [statistical method as in outcome 1, analysis 1]; t-statistic = -4.87 — t-statistic associated with the contrast of the MMRM model for dose-response pattern 2. Lower value indicates pattern provides better fit to data
Statistical Analysis 6: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.0021, MMRM — p-value (adjusted to control Type I error in multiple testing) for dose-response pattern 3 (Placebo=2.5 mg=5.0 mg<10.0 mg); [statistical method as in outcome 1, analysis 1]; t-statistic = -3.40 — t-statistic associated with the contrast of the MMRM model for dose-response pattern 3. Lower value indicates pattern provides better fit to data
Statistical Analysis 7: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.0001, MMRM — p-value (adjusted to control Type I error in multiple testing) for dose-response pattern 4 (Placebo<2.5 mg<5.0 mg<10.0 mg); [statistical method as in outcome 1, analysis 1]; t-statistic = -5.28 — t-statistic associated with the contrast of the MMRM model for dose-response pattern 4. Lower value indicates pattern provides better fit to data
Statistical Analysis 8: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.0001, MMRM — p-value (adjusted to control Type I error in multiple testing) for dose-response pattern 5 (Placebo=2.5 mg<5.0 mg<10.0 mg); [statistical method as in outcome 1, analysis 1]; t-statistic = -4.64 — t-statistic associated with the contrast of the MMRM model for dose-response pattern 5. Lower value indicates pattern provides better fit to data
Statistical Analysis 9: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.0001, MMRM — p-value (adjusted to control Type I error in multiple testing) for dose-response pattern 6 (Placebo<2.5 mg=5.0 mg<10.0 mg); [statistical method as in outcome 1, analysis 1]; t-statistic = -5.07 — t-statistic associated with the contrast of the MMRM model for dose-response pattern 6. Lower value indicates pattern provides better fit to data
Statistical Analysis 10: Comparison: Placebo vs Asenapine 2.5 mg BID vs Asenapine 5.0 mg BID vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.0001, MMRM — p-value (adjusted to control Type I error in multiple testing) for dose-response pattern 7 (Placebo<2.5 mg<5.0 mg=10.0 mg); [statistical method as in outcome 1, analysis 1]; t-statistic = -5.49 — t-statistic associated with the contrast of the MMRM model for dose-response pattern 7. Lower value indicates pattern provides better fit to data

2. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale for Use in Bipolar Disorder (CGI-BP) Overall Score at Day 21
Description: Change from baseline in CGI-BP overall score at Day 21 is the Key Secondary Outcome Measure. The CGI-BP is a clinician-rated instrument for assessing bipolar illness that includes subscales assessing mania and depression. This measure reports one item within the CGI-BP, which is a 7-point scale assessing the severity of the participant's overall bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 21; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 21
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 21 value of CGI-BP overall score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 79 | 88 | 87 | 81
score on a scale | -0.7 (0.9) | -1.3 (1.1) | -1.4 (1.0) | -1.4 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM — p-value is adjusted by Hochberg's method for testing three asenapine groups versus the placebo group; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.6, 95% CI 2-sided [-0.9 to -0.3] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM — p-value is adjusted by Hochberg's method for testing three asenapine groups versus the placebo group; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.7, 95% CI 2-sided [-0.9 to -0.4] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM — p-value is adjusted by Hochberg's method for testing three asenapine groups versus the placebo group; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.7, 95% CI 2-sided [-1.0 to -0.4] — Estimate is asenapine versus placebo

3. Secondary Outcome: Total Y-MRS 50% Responders at Days 4, 7, 14 and 21
Description: A total Y-MRS 50% responder was defined as a participant who had a reduction from baseline to the identified study visit of at least 50% in the Y-MRS total score. The Y-MRS is an 11-item clinician-rated instrument for assessing the severity of manic episodes. A severity rating is assigned to each of the 11 items, based on the participant's subjective report of his or her condition over the previous 48 hours and the clinician's observations during the interview, with the emphasis on the latter. The Y-MRS total score for each participant is the sum of the ratings for the 11 individual items, and can range from 0-60 with higher scores indicating greater severity of symptoms. This analysis used a Last-Observation-Carried-Forward (LOCF) approach; if at a given visit no Y-MRS total score was available for determining whether a participant was a responder, the last available post-baseline on-treatment assessment prior to that visit was used.
Time Frame: Baseline and Days 4, 7, 14 and 21
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included for a visit, a Y-MRS total score must be available for that visit or a prior post-baseline on-treatment visit
Measure: Number; unit: participants
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 98 | 101 | 98 | 98
participants
  Day 4 (n=95, 98, 93, 90) | 7 | 19 | 20 | 13
  Day 7 (n=98, 101, 98, 98) | 14 | 33 | 31 | 37
  Day 14 (n=98, 101, 98, 98) | 20 | 36 | 50 | 50
  Day 21 (n=98, 101, 98, 98) | 27 | 42 | 53 | 51
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Analysis is for asenapine versus placebo on Day 4 (LOCF); Test type: Superiority or Other; p = 0.018, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 3.0, 95% CI 2-sided [1.2 to 7.6] — OR was adjusted for baseline. An OR of >1 is considered to mean that asenapine has a higher probability of achieving Total Y-MRS 50% response
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Analysis is for asenapine versus placebo on Day 4 (LOCF); Test type: Superiority or Other; p = 0.008, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 3.4, 95% CI 2-sided [1.4 to 8.6] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; Analysis is for asenapine versus placebo on Day 4 (LOCF); Test type: Superiority or Other; p = 0.129, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 2.1, 95% CI 2-sided [0.8 to 5.6] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Asenapine 2.5 mg BID; Analysis is for asenapine versus placebo on Day 7 (LOCF); Test type: Superiority or Other; p = 0.003, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.4 to 5.9] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Asenapine 5.0 mg BID; Analysis is for asenapine versus placebo on Day 7 (LOCF); Test type: Superiority or Other; p = 0.005, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 2.8, 95% CI 2-sided [1.4 to 5.6] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Asenapine 10.0 mg BID; Analysis is for asenapine versus placebo on Day 7 (LOCF); Test type: Superiority or Other; p < 0.001, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 3.6, 95% CI 2-sided [1.8 to 7.3] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Asenapine 2.5 mg BID; Analysis is for asenapine versus placebo on Day 14 (LOCF); Test type: Superiority or Other; p = 0.018, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 2.2, 95% CI 2-sided [1.1 to 4.1] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Asenapine 5.0 mg BID; Analysis is for asenapine versus placebo on Day 14 (LOCF); Test type: Superiority or Other; p < 0.001, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 4.1, 95% CI 2-sided [2.2 to 7.6] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs Asenapine 10.0 mg BID; Analysis is for asenapine versus placebo on Day 14 (LOCF); Test type: Superiority or Other; p < 0.001, Regression, Logistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 4.1, 95% CI 2-sided [2.2 to 7.6] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs Asenapine 2.5 mg BID; Analysis is for asenapine versus placebo on Day 21 (LOCF); Test type: Superiority or Other; p = 0.042, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.0 to 3.4] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs Asenapine 5.0 mg BID; Analysis is for asenapine versus placebo on Day 21 (LOCF); Test type: Superiority or Other; p < 0.001, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 3.2, 95% CI 2-sided [1.7 to 5.8] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs Asenapine 10.0 mg BID; Analysis is for asenapine versus placebo on Day 21 (LOCF); Test type: Superiority or Other; p < 0.001, Regression, Logistic — 95% Confidence Interval and p-value are based on Wald statistic; Model included terms of treatment and baseline Y-MRS total score; Odds Ratio (OR) = 2.9, 95% CI [1.6 to 5.3] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in CGI-BP Mania Score at Day 4
Description: The CGI-BP is a clinician-rated instrument for assessing bipolar illness that includes subscales assessing mania and depression. This measure reports one item within the CGI-BP, which is a 7-point scale assessing the severity of the mania component of the participant's bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 4; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 4
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 4 value of CGI-BP mania score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 93 | 97 | 93 | 90
score on a scale | -0.3 (0.6) | -0.6 (0.8) | -0.5 (0.7) | -0.5 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.014, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.25, 95% CI 2-sided [-0.45 to -0.05] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.107, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.17, 95% CI 2-sided [-0.37 to 0.04] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.039, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.21, 95% CI 2-sided [-0.42 to -0.01] — Estimate is asenapine versus placebo

5. Secondary Outcome: Change From Baseline in CGI-BP Mania Score at Day 7
Description: The CGI-BP is a clinician-rated instrument for assessing bipolar illness that includes subscales assessing mania and depression. This measure reports one item within the CGI-BP, which is a 7-point scale assessing the severity of the mania component of the participant's bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 7; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 7
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 7 value of CGI-BP mania score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 95 | 98 | 95 | 97
score on a scale | -0.5 (0.7) | -0.9 (0.9) | -0.9 (1.0) | -0.9 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.006, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.33, 95% CI 2-sided [-0.56 to -0.10] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.35, 95% CI 2-sided [-0.59 to -0.12] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.44, 95% CI 2-sided [-0.67 to -0.21] — Estimate is asenapine versus placebo

6. Secondary Outcome: Change From Baseline in CGI-BP Mania Score at Day 14
Description: The CGI-BP is a clinician-rated instrument for assessing bipolar illness that includes subscales assessing mania and depression. This measure reports one item within the CGI-BP, which is a 7-point scale assessing the severity of the mania component of the participant's bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 14; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 14
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 14 value of CGI-BP mania score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 89 | 91 | 90 | 91
score on a scale | -0.6 (1.0) | -1.1 (1.0) | -1.4 (1.0) | -1.3 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.011, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.34, 95% CI 2-sided [-0.61 to -0.08] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.63, 95% CI 2-sided [-0.89 to -0.36] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.61, 95% CI 2-sided [-0.88 to -0.35] — Estimate is asenapine versus placebo

7. Secondary Outcome: Change From Baseline in CGI-BP Mania Score at Day 21
Description: The CGI-BP is a clinician-rated instrument for assessing bipolar illness that includes subscales assessing mania and depression. This measure reports one item within the CGI-BP, which is a 7-point scale assessing the severity of the mania component of the participant's bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 21; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 21
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 21 value of CGI-BP mania score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 79 | 88 | 87 | 81
score on a scale | -0.7 (0.9) | -1.3 (1.1) | -1.5 (1.1) | -1.4 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.61, 95% CI 2-sided [-0.90 to -0.32] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.75, 95% CI 2-sided [-1.04 to -0.46] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.74, 95% CI 2-sided [-1.03 to -0.45] — Estimate is asenapine versus placebo

8. Secondary Outcome: Change From Baseline in CGI-BP Depression Score at Day 4
Description: The CGI-BP is a clinician-rated instrument for assessing bipolar illness that includes subscales assessing mania and depression. This measure reports one item within the CGI-BP, which is a 7-point scale assessing the severity of the depression component of the participant's bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 4; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 4
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 4 value of CGI-BP depression score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 92 | 97 | 93 | 90
score on a scale | -0.2 (0.7) | -0.3 (0.8) | -0.2 (1.0) | -0.1 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.536, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.07, 95% CI 2-sided [-0.28 to 0.15] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.811, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.03, 95% CI 2-sided [-0.24 to 0.19] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.556, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = 0.07, 95% CI 2-sided [-0.15 to 0.28] — Estimate is asenapine versus placebo

9. Secondary Outcome: Change From Baseline in CGI-BP Depression Score at Day 7
Description: The CGI-BP is a clinician-rated instrument for assessing bipolar illness that includes subscales assessing mania and depression. This measure reports one item within the CGI-BP, which is a 7-point scale assessing the severity of the depression component of the participant's bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 7; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 7
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 7 value of CGI-BP depression score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 94 | 98 | 95 | 97
score on a scale | -0.4 (0.9) | -0.5 (0.8) | -0.5 (1.1) | -0.5 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.053, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.21, 95% CI 2-sided [-0.42 to 0.00] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.094, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.18, 95% CI 2-sided [-0.40 to 0.03] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.178, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.15, 95% CI 2-sided [-0.36 to 0.07] — Estimate is asenapine versus placebo

10. Secondary Outcome: Change From Baseline in CGI-BP Depression Score at Day 14
Description: The CGI-BP is a clinician-rated instrument for assessing bipolar illness that includes subscales assessing mania and depression. This measure reports one item within the CGI-BP, which is a 7-point scale assessing the severity of the depression component of the participant's bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 14; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 14
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 14 value of CGI-BP depression score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 88 | 91 | 90 | 91
score on a scale | -0.5 (1.1) | -0.5 (1.0) | -0.7 (1.0) | -0.6 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.506, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.08, 95% CI 2-sided [-0.33 to 0.16] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.131, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.19, 95% CI 2-sided [-0.43 to 0.06] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.211, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.16, 95% CI 2-sided [-0.40 to 0.09] — Estimate is asenapine versus placebo

11. Secondary Outcome: Change From Baseline in CGI-BP Depression Score at Day 21
Description: The CGI-BP is a clinician-rated instrument for assessing bipolar illness that includes subscales assessing mania and depression. This measure reports one item within the CGI-BP, which is a 7-point scale assessing the severity of the depression component of the participant's bipolar illness, with ratings from 1=normal, not ill to 7=very severely ill. The reported measure is the change from baseline at Day 21; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 21
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 21 value of CGI-BP depression score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 78 | 88 | 87 | 81
score on a scale | -0.4 (1.0) | -0.6 (1.1) | -0.8 (1.1) | -0.6 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.079, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.23, 95% CI 2-sided [-0.49 to 0.03] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.010, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.34, 95% CI 2-sided [-0.60 to -0.08] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.139, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.20, 95% CI 2-sided [-0.46 to 0.06] — Estimate is asenapine versus placebo

12. Secondary Outcome: Change From Baseline in Children's Depression Rating Scale, Revised (CDRS-R) Total Score at Day 7
Description: The CDRS-R is a 17-item clinician-rated instrument for assessing the presence and severity of depressive symptoms in children. Fourteen of the 17 items are rated on a scale of 1-7 and 3 of the items are rated on a scale of 1-5, with higher scores indicating greater severity of symptoms. The CDRS-R total score for each participant is the sum of the ratings for the 17 individual items, and can range from 17-113, with higher scores indicating greater severity of symptoms. The reported measure is the change from baseline at Day 7; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 7
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 7 value of CDRS-R total score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 94 | 95 | 91 | 95
score on a scale | -4.1 (8.1) | -6.1 (7.1) | -6.1 (8.0) | -5.9 (8.5)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -2.61, 95% CI 2-sided [-4.38 to -0.83] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.017, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -2.17, 95% CI 2-sided [-3.95 to -0.39] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.017, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -2.16, 95% CI 2-sided [-3.93 to -0.38] — Estimate is asenapine versus placebo

13. Secondary Outcome: Change From Baseline in CDRS-R Total Score at Day 14
Description: The CDRS-R is a 17-item clinician-rated instrument for assessing the presence and severity of depressive symptoms in children. Fourteen of the 17 items are rated on a scale of 1-7 and 3 of the items are rated on a scale of 1-5, with higher scores indicating greater severity of symptoms. The CDRS-R total score for each participant is the sum of the ratings for the 17 individual items, and can range from 17-113, with higher scores indicating greater severity of symptoms. The reported measure is the change from baseline at Day 14; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 14
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 14 value of CDRS-R total score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 88 | 89 | 90 | 90
score on a scale | -5.5 (8.1) | -5.8 (6.5) | -8.7 (10.5) | -6.6 (8.8)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.395, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -0.79, 95% CI 2-sided [-2.62 to 1.04] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.009, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -2.44, 95% CI 2-sided [-4.26 to -0.63] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.121, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.44, 95% CI 2-sided [-3.27 to 0.38] — Estimate is asenapine versus placebo

14. Secondary Outcome: Change From Baseline in CDRS-R Total Score at Day 21
Description: The CDRS-R is a 17-item clinician-rated instrument for assessing the presence and severity of depressive symptoms in children. Fourteen of the 17 items are rated on a scale of 1-7 and 3 of the items are rated on a scale of 1-5, with higher scores indicating greater severity of symptoms. The CDRS-R total score for each participant is the sum of the ratings for the 17 individual items, and can range from 17-113, with higher scores indicating greater severity of symptoms. The reported measure is the change from baseline at Day 21; improvement in symptoms is represented by negative values.
Time Frame: Baseline and Day 21
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and an on-treatment Day 21 value of CDRS-R total score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 78 | 87 | 87 | 81
score on a scale | -6.1 (8.8) | -6.9 (7.3) | -8.7 (11.4) | -6.8 (8.9)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.135, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.44, 95% CI 2-sided [-3.33 to 0.45] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.023, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -2.19, 95% CI 2-sided [-4.08 to -0.30] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.189, MMRM; [statistical method as in outcome 1, analysis 1]; Difference in LS Means = -1.28, 95% CI 2-sided [-3.20 to 0.63] — Estimate is asenapine versus placebo

15. Secondary Outcome: Change From Baseline in Children's Global Assessment Scale (CGAS) Score at Day 21
Description: CGAS is a 100-point scale measuring psychological, social, and school functioning in children aged 6-17. Minimum scores ranged from 1-10, representing the need for constant supervision (worse result) to maximum scores of 91-100, representing superior functioning (better result). The reported measure is the change from baseline at Day 21; improvement in functioning is represented by positive values. This analysis used an LOCF approach; if no Day 21 value was available for a participant, the last available post-baseline on-treatment assessment prior to the Day 21 assessment was used.
Time Frame: Baseline and Day 21
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and at least 1 post-baseline on-treatment value of CGAS score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 84 | 93 | 91 | 85
score on a scale | 6.0 (8.1) | 9.4 (9.5) | 13.0 (11.6) | 10.8 (9.7)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Test type: Superiority or Other; p = 0.002, ANCOVA; Model included terms of (pooled) site, treatment and baseline; Difference in LS Means = 4.29, 95% CI 2-sided [1.56 to 7.02] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Model included terms of (pooled) site, treatment and baseline; Difference in LS Means = 6.95, 95% CI 2-sided [4.22 to 9.68] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; Test type: Superiority or Other; p < 0.001, ANCOVA; Model included terms of (pooled) site, treatment and baseline; Difference in LS Means = 5.11, 95% CI 2-sided [2.31 to 7.91] — Estimate is asenapine versus placebo

16. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) Total Score at Day 21
Description: PQ-LES-Q is a questionnaire to assess quality of life enjoyment and satisfaction in children and adolescents. The participant is asked to rate 15 items reflecting quality of life with respect to the previous week on a scale of 1=very poor to 5=very good. Items 1-14 assess specific areas (e.g., your health, your mood or feelings); Item 15 is a global assessment of overall quality of life. The PQ-LES-Q total score for each participant was calculated as the sum of the rating assigned to each of the first 14 items, and ranged from 14 to 70 with a higher score indicating better quality of life. The reported measure is the change from baseline at Day 21; improvement in quality of life is represented by positive values. This analysis used an LOCF approach; if no Day 21 value was available for a participant, the last available post-baseline on-treatment assessment prior to the Day 21 assessment was used.
Time Frame: Baseline and Day 21
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and at least 1 post-baseline on-treatment value of PQ-LES-Q total score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 84 | 92 | 90 | 84
score on a scale | 1.5 (8.2) | 3.7 (8.6) | 2.5 (10.8) | 4.0 (9.8)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Test type: Superiority or Other; p = 0.050, ANCOVA; Model included terms of (pooled) site, treatment and baseline; Difference in LS Means = 2.24, 95% CI 2-sided [-0.00 to 4.48] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p = 0.239, ANCOVA; Model included terms of (pooled) site, treatment and baseline; Difference in LS Means = 1.35, 95% CI 2-sided [-0.90 to 3.59] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; Test type: Superiority or Other; p = 0.018, ANCOVA; Model included terms of (pooled) site, treatment and baseline; Difference in LS Means = 2.78, 95% CI 2-sided [0.48 to 5.08] — Estimate is asenapine versus placebo

17. Secondary Outcome: Change From Baseline in PQ-LES-Q Overall Score (i.e., Item 15) at Day 21
Description: PQ-LES-Q is a questionnaire to assess quality of life enjoyment and satisfaction in children and adolescents. The participant is asked to rate 15 items reflecting quality of life with respect to the previous week on a scale of 1=very poor to 5=very good. Items 1-14 assess specific areas (e.g., your health, your mood or feelings); Item 15 is a global assessment of overall quality of life. The Item 15 result is defined to be the PQ-LES-Q overall score, and ranged from 1 to 5 with a higher score indicating better quality of life. The reported measure is the change from baseline at Day 21; improvement in quality of life is represented by positive values. This analysis used an LOCF approach; if no Day 21 value was available for a participant, the last available post-baseline on-treatment assessment prior to the Day 21 assessment was used.
Time Frame: Baseline and Day 21
Population: Randomized participants who received at least 1 dose of study drug and had both a baseline and at least 1 post-baseline on-treatment Y-MRS total score (this group is termed the efficacy FAS); also, to be included a baseline and at least 1 post-baseline on-treatment value of PQ-LES-Q overall score must be available for a participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Number analyzed (Participants) | 84 | 92 | 90 | 84
score on a scale | -0.0 (0.9) | 0.4 (1.0) | 0.1 (1.0) | 0.2 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Asenapine 2.5 mg BID; Test type: Superiority or Other; p = 0.001, ANCOVA; Model included terms of (pooled) site, treatment and baseline; Difference in LS Means = 0.39, 95% CI 2-sided [0.15 to 0.62] — Estimate is asenapine versus placebo
Statistical Analysis 2: Comparison: Placebo vs Asenapine 5.0 mg BID; Test type: Superiority or Other; p = 0.135, ANCOVA; Model included terms of (pooled) site, treatment and baseline; Difference in LS Means = 0.18, 95% CI 2-sided [-0.06 to 0.41] — Estimate is asenapine versus placebo
Statistical Analysis 3: Comparison: Placebo vs Asenapine 10.0 mg BID; Test type: Superiority or Other; p = 0.044, ANCOVA; Model included terms of (pooled) site, treatment and baseline; Difference in LS Means = 0.25, 95% CI 2-sided [0.01 to 0.49] — Estimate is asenapine versus placebo

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study drug (Up to 51 days)
Arm/Group | Placebo | Asenapine 2.5 mg BID | Asenapine 5.0 mg BID | Asenapine 10.0 mg BID
Serious Adverse Events (participants affected / at risk) | 3/101 | 0/104 | 2/99 | 2/99
Other Adverse Events (participants affected / at risk) | 30/101 | 68/104 | 70/99 | 72/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Asenapine 2.5 mg BID (N=104) | Asenapine 5.0 mg BID (N=99) | Asenapine 10.0 mg BID (N=99)
BIPOLAR DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BIPOLAR I DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
MANIA (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUICIDAL BEHAVIOUR (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Asenapine 2.5 mg BID (N=104) | Asenapine 5.0 mg BID (N=99) | Asenapine 10.0 mg BID (N=99)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 (6) | 5 (5) | 2 (2) | 3 (3)
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 2 (2) | 18 (18) | 18 (19) | 20 (21)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 6 (6) | 6 (6) | 6 (7)
PARAESTHESIA ORAL (Gastrointestinal disorders) | 2 (2) | 9 (9) | 9 (9) | 11 (11)
FATIGUE (General disorders) | 5 (5) | 4 (4) | 8 (8) | 13 (13)
WEIGHT INCREASED (Investigations) | 0 (0) | 6 (6) | 2 (2) | 2 (2)
INCREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 10 (10) | 9 (10) | 6 (6)
DIZZINESS (Nervous system disorders) | 3 (4) | 6 (6) | 10 (11) | 5 (5)
DYSGEUSIA (Nervous system disorders) | 2 (2) | 4 (4) | 5 (5) | 9 (9)
HEADACHE (Nervous system disorders) | 6 (6) | 8 (11) | 11 (12) | 9 (10)
SEDATION (Nervous system disorders) | 5 (5) | 16 (16) | 19 (19) | 18 (20)
SOMNOLENCE (Nervous system disorders) | 6 (6) | 34 (39) | 34 (36) | 31 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is planned to first publish/present trial results together with the other sites, unless permission is obtained from Sponsor to publish separate results. Sponsor must be able to review all proposed results communications regarding study 45 days prior to submission for publication/presentation. If there is disagreement concerning appropriateness of the materials, Investigator and Sponsor must meet to make a good faith effort to discuss/resolve disagreement prior to submission for publication.